CLINICAL TRIAL: NCT00623961
Title: Validation Study of Positive Phenomena in Neuropathic Pain
Brief Title: Validation Study of Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0425
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Neuropathic Pain From Spinal Cord Injury; Diabetic Peripheral Neuropathy; Post Herpetic Pain
Keywords: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to validate clinically evoked or obtained objective pain signs with the patient's corresponding quantified subjective pain symptoms. This will allow for validation of objective clinical pain signs to then be used to begin to classify patients with pain based on symptoms and signs. This then can be used as a basis for further study of neuropathic pain mechanisms in human patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age and older, and able to provide informed consent and communicate in English. Pain rating inclusion criteria will be pain greater than 3 up to 9, as rated on the 0-10 pain scale, where 10 is the worst pain imaginable. This rating is based on the numeric pain rating scale (NPRS).
* PHN - Subjects with PHN will have a history of pain of at least 6 months duration in the area that was the site of a zoster rash resulting in nerve injury. In most cases, subjects experience a number of sensory abnormalities in the affected area, ranging from pain to numbness, and various degrees of hypersensitivity. Subjects with PHN must otherwise be in stable health. Pain rating inclusion criteria for PHN subjects will be pain greater than 3 up to 9, as rated on the 0-10 pain scale, where 10 is the worst pain imaginable.
* PDN - Subjects with diabetes mellitus and neuropathy who have a history of pain, predominantly in the lower extremities, of at least 6 months duration qualify for the diagnosis of PDN for purposes of this study. In most cases PDN is due to small fiber neuropathy, so physical examination should yield sensory abnormalities, such as pain, paresthesiae and numbness. Motor function and stretch reflex abnormalities are common but not necessary for inclusion. PDN patients in whom large fiber functions are affected, experience weakness and decreased or absent stretch reflexes, respectively, and are eligible for this study. Other causes of neuropathy will be excluded. PDN patients with pain rating of greater than 3 up to 9 on 0-10 scale will be included.
* SCI pain - Subjects with SCI and pain of at least 6 months duration will be invited to participate. In most cases, these subjects' sensory, motor and stretch reflex abnormalities are consistent with SCI. Sensory findings range form complete loss of sensation to preservation of all sensory modalities. Motor findings range from mild weakness to complete paralysis. Stretch reflexes are most frequently increased though in a few patients they can be absent. Based on the constellation of sensory and motor findings in particular patients, diagnosis of complete versus incomplete SCI is made. In this study we will study patients with incomplete SCI who have pain at level of injury or below level of injury, or both. Subjects with SCI who have pain rating of greater than 3 up to 9 on 0-10 scale will be included.

Exclusion Criteria:

* Patients with pain due to disorders other than PDN, PTN, or SCI, as well as unknown causes, will be excluded.
* Patients with neuropathies from causes such as vasculitis, demyelinating polyneuropathies, HIV-associated neuropathy, and paraneoplastic and post-infectious neuropathies will be excluded.
* Patients with chemotherapy-induced neuropathy will be excluded.
* Patients who suffer from pain due to different pain mechanisms will be excluded.
* Patients with other pain (at a different site) that is more severe than their PDN or PTN pain will be excluded.
* Patients with a history of recent or ongoing alcohol or other drug addiction disorders (as self-reported or previously documented in the medical record) will be excluded.
* Patients who are determined to have cognitive and reading impairments which would preclude them from completing questionnaires will be excluded.
* Patients whose chronic medical and psychiatric comorbidities are not under optimal control, or who are currently experiencing an acute exacerbation of a medical or psychiatric comorbidity, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic pain from the following diagnosis groups: post-herperic neuralgia, painful diabetic neuropathy, and spinal cord injury will be included in the study if their pain is of at least 6 months duration.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Validation of neuropathic pain sensory sign and corresponding symptoms | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Backonja, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospitals and Clinics, Madison, Wisconsin, United States